CLINICAL TRIAL: NCT05010512
Title: Clinical Performance of Two Commercial, Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLU484-P002
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Refractive Errors; Ametropia; Myopia
Keywords: Contact lenses
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DT1, then Infuse (Other): Delefilcon A contact lenses worn first, with kalifilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 (-0/+3) days on a daily wear, daily disposable basis.
  Interventions: Device: Delefilcon A contact lenses; Device: Kalifilcon A contact lenses
- Infuse, then DT1 (Other): Kalifilcon A contact lenses worn first, with delefilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 (-0/+3) days on a daily wear, daily disposable basis.
  Interventions: Device: Delefilcon A contact lenses; Device: Kalifilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Commercially available silicone hydrogel contact lenses used as indicated
  Other Names: DAILIES TOTAL1®; DT1
Device: Kalifilcon A contact lenses — Commercially available silicone hydrogel contact lenses used as indicated
  Other Names: Bausch + Lomb INFUSE™; Infuse

SUMMARY:
The purpose of this study is to compare the clinical performance of DAILIES TOTAL1 ( DT1) contact lenses with Infuse contact lenses.

DETAILED DESCRIPTION:
Subjects will wear two products and be expected to attend 3 office visits. The individual duration of participation will be approximately 3 weeks, which includes 16 to 22 days of lens wear.

ELIGIBILITY:
Key Inclusion Criteria:

* Habitually wears soft contact lenses in both eyes at least 5 days per week and at least 10 hours per day;
* At least 3 months of contact lens wearing experience;
* Less than or equal to 0.75 diopter (D) astigmatism in each eye;
* Best Corrected Visual Acuity (BCVA) better than or equal to 20/25 in each eye.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Current/previous DAILIES TOTAL1 and/or Infuse habitual lens wearer;
* Monovision and/or multifocal lens wearer;
* Routinely sleeps in habitual contact lenses.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Alcon Investigator 6355, Orlando, Florida
  - Alcon Investigator 6418, Tallahassee, Florida
  - Alcon Investigator 3950, Bloomington, Illinois
  - Alcon Investigator 6614, Franklin Park, Illinois
  - Alcon Investigator 6583, Eden Prairie, Minnesota
  - Alcon Investigator 3382, Wyomissing, Pennsylvania
  - Alcon Investigator 6353, Memphis, Tennessee
  - Alcon Investigator 2786, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 investigative sites in the United States.
Pre-assignment Details: Of the 112 enrolled, one subject was exited prior to randomization as a screen failure. This reporting group includes all randomized subjects (111).
Groups:
- DT1, Then Infuse: Delefilcon A contact lenses worn first, with kalifilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 (-0/+3) days on a daily wear, daily disposable basis.
- Infuse, Then DT1: Kalifilcon A contact lenses worn first, with delefilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 (-0/+3) days on a daily wear, daily disposable basis.
Period: Period 1, 8 (-0/+3) Days
Arm/Group | DT1, Then Infuse | Infuse, Then DT1
Started | 55 | 56
Completed | 55 | 56
Not Completed | 0 | 0
Period: Period 2, 8 (-0/+3) Days
Arm/Group | DT1, Then Infuse | Infuse, Then DT1
Started | 55 | 56
Completed | 55 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized subjects exposed to any study lenses evaluated in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | DT1, Then Infuse | Infuse, Then DT1 | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (8.2) | 32.4 (7.4) | 33.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 77
  Male | 14 | 20 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 49 | 53 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 52 | 102
  Black or African American | 4 | 3 | 7
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 1 | 1
  Multi-racial | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 55 | 56 | 111

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance VA (logMAR) With Study Lenses
Description: Distance visual acuity (VA) was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 8 (-0/+3), each study lens type
Population: FAS with non-missing response (eye)
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- DT1 (Delefilcon A): Delefilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 (-0/+3) days on a daily wear, daily disposable basis
- Infuse (Kalifilcon A): Kalifilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 (-0/+3) days on a daily wear, daily disposable basis
Arm/Group | DT1 (Delefilcon A) | Infuse (Kalifilcon A)
Number analyzed (Participants) | 111 | 110
Number analyzed (eyes) | 222 | 220
logMAR | -0.10 (0.006) | -0.10 (0.006)
Statistical Analysis 1: Comparison: DT1 (Delefilcon A) vs Infuse (Kalifilcon A); Test type: Non-Inferiority — Noninferiority in distance VA was declared if the least squares means difference upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least Squares Mean Difference = -0.00, 95% CI 1-sided [upper limit 0.01], Standard Error of Mean 0.004 — LSM results based on mixed effects repeated measures model with terms for lens, period and sequence as fixed effects, subject as a random effect. Difference = DT1 minus Infuse

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, 16-22 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- DT1 Ocular; DT1 Nonocular: Events reported in this group occurred while exposed to the delefilcon A contact lenses
- Infuse Ocular; Infuse Nonocular: Events reported in this group occurred while exposed to the kalifilcon A contact lenses
Arm/Group | Pretreatment | DT1 Ocular | DT1 Nonocular | Infuse Ocular | Infuse Nonocular
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/222 | 0/111 | 0/222 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/222 | 0/111 | 0/222 | 0/111
Other Adverse Events (participants affected / at risk) | 0/111 | 0/222 | 0/111 | 0/222 | 0/111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT05010512/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT05010512/SAP_001.pdf